CLINICAL TRIAL: NCT05593744
Title: Study on the Correlation Between Thyroid Dysfunction Induced by Anti PD-1 Therapy and Prognosis in Patients With Advanced Carcinoma
Brief Title: Thyroid Dysfunction Induced by Anti-PD-1 Therapy in Patients With Advanced Carcinoma
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: SDU-KYLL-202208-042
Record Dates: First submitted 2022-10-18; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroid dysfunction: Patients had thyroid dysfunction during anti-PD-1 therapy.
  Interventions: Other: no intervention
- No thyroid dysfunction: Patients didn't have thyroid dysfunction during anti-PD-1 therapy.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observational study so not involved intervention

SUMMARY:
In this study, we monitored patients with advanced malignant tumors who received anti-PD-1 therapy to observe the characteristic of anti-PD-1 therapy-induced thyroid dysfunction and its correlation with prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years or older
* Confirmed diagnosis of malignancy
* Received anti-PD-1 therapy

Exclusion Criteria:

* Thyroid malignancy or history of thyroid malignancy
* Thyroid dysfunction before anti-PD-1 therapies
* Previous ICIs treatment
* Less than 2 cycles of anti-PD-1 treatment
* No thyroid function monitoring during treatment
* Known pituitary disease
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced carcinoma who received anti-PD-1 therapy at East Branch of Qilu Hospital of Shandong University
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Through study completion, an average of 17 weeks
  The time between initiation of anti-PD-1 therapy and disease progression or death, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Y, Li Q, Xu L, Zheng Y, Wang Y, Liu Y, Zhang R, Liao L, Dong J. Thyroid dysfunction induced by anti-PD-1 therapy is associated with a better progression-free survival in patients with advanced carcinoma. J Cancer Res Clin Oncol. 2023 Dec;149(18):16501-16510. doi: 10.1007/s00432-023-05364-z. Epub 2023 Sep 15. PMID 37715029